CLINICAL TRIAL: NCT01584050
Title: Relative Bioavailability of Folic Acid and L-5-Methlytetrahydrofolate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: H10-03426
Record Dates: First submitted 2012-04-20; First posted 2012-04-24 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Vitamin B12 Deficiency
MeSH Terms: conditions — Vitamin B 12 Deficiency | interventions — 5-methyltetrahydrofolate; levomefolate calcium; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- L-MTHF (Active Comparator)
  Interventions: Dietary Supplement: L-5-methyltetrahydrofolate (Metafolin ®)
- folic acid (Active Comparator)
  Interventions: Dietary Supplement: folic acid
- placebo (methyl cellulose) (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-5-methyltetrahydrofolate (Metafolin ®) — dosage: 1000 μg, frequency: once daily, duration: 12 weeks
  Arms: L-MTHF
Dietary Supplement: folic acid — dosage: 1000 μg, frequency: once daily, duration: 12 weeks
  Arms: folic acid
Dietary Supplement: Placebo — frequency: once daily, duration: 12 weeks
  Arms: placebo (methyl cellulose)

SUMMARY:
Folic acid, a form of the vitamin folate, is added to grain products in Canada to help reduce birth defects. Folic acid is the synthetic form of folate and is very stable (doesn't break down) when added to foods. There are emerging health concerns about chronic folic acid consumption. Recently another more natural form of folate, L-5-methyltetrahydrofolate (L-MTHF) has become available. The investigators plan to conduct a randomized trial in women to determine if supplements containing L-MTHF consumed over three months raises blood folate levels as much as supplements containing folic acid. The investigators hypothesize that L-MTHF will increase red cell folate over 12 weeks to same extent as equimolar folic acid.

DETAILED DESCRIPTION:
The proposed study is a twelve week, cross-sectional, double blind, randomized controlled trial. The sample population will consist of one-hundred fifty healthy adult volunteers. All participants will be Malaysian women between eighteen and forty-two years of age. Study participants will be recruited by word of mouth and through advertisements placed in hospitals and universities starting in January 2011. Study participants will be randomly assigned to 1 of 3 treatment groups: 1) 1000ug L-MTHF 2) 1000ug folic acid 3) placebo (methyl cellulose). All treatments will be given in capsule form. Blood samples will be collected at baseline, 6 and 12 weeks.

The primary outcome measure is red cell folate. A sample size of 45 subjects per group will allow us to detect a minimum difference of 100 nmol/L red cell folate assuming an alpha 0.05, a beta of 0.8 a SD of 183 nmol/L. Accounting for a 10% attrition rate we will enroll 50 women per group. The study will be analyzed as intent to treat. Baseline characteristics and compliance between treatment groups will be compared using a one-way ANOVA for continuous variables and chi-square analyses for categorical variables. The difference in measurements between the treatment groups at week 12 will be determined by regression analysis, controlling for baseline values.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian nationality

Exclusion Criteria:

* Pregnancy
* Vitamin supplement users
* Chronic disease
* prior neural tube defect affected pregnancy

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Red cell folate (nmol/L) | 12 weeks
  Measured at baseline, 6 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tim Green, PhD, Principal Investigator — University of British Columbia
Locations (2):
- University of British Columbia, Vancouver, British Columbia, Canada
- Universiti Putra Malaysia, Serdang, Selangor, Malaysia

REFERENCES:
- [Derived] Henderson AM, Aleliunas RE, Loh SP, Khor GL, Harvey-Leeson S, Glier MB, Kitts DD, Green TJ, Devlin AM. l-5-Methyltetrahydrofolate Supplementation Increases Blood Folate Concentrations to a Greater Extent than Folic Acid Supplementation in Malaysian Women. J Nutr. 2018 Jun 1;148(6):885-890. doi: 10.1093/jn/nxy057. PMID 29878267